CLINICAL TRIAL: NCT01866709
Title: A Phase 4, Single-center, Prospective, Double-blind, Placebo-controlled, Randomized Study to Investigate the Safety and Efficacy of Sodium Polystyrene Sulfonate (SPS) in Subjects With Hyperkalemia.
Brief Title: Safety and Efficacy of Sodium Polystyrene Sulfonate in Hyperkalemia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Risk/benefit determination showed study revealed negative safety issues.
Sponsor: ZS Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SPS-001
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Results first posted 2014-09-03 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Hyperkalemia
MeSH Terms: conditions — Hyperkalemia | interventions — polystyrene sulfonic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium Polystyrene Sulfonate (Active Comparator): Oral suspension in water of 15g sodium polystyrene sulfonate administered three times (tid) daily for 48 hours without co-administration of Sorbitol.
  Interventions: Drug: Sodium polystyrene sulfonate
- Silicified microcrystalline cellulose (Placebo Comparator): Oral suspension of placebo blended with pigment to have the same appearance, taste, odor and mode of administration as SPS.
  Interventions: Drug: Silicified microcrystalline cellulose

INTERVENTIONS:
Drug: Sodium polystyrene sulfonate — Oral suspension in water of 15g sodium polystyrene sulfonate administered three times (tid) daily for 48 hours without co-administration of Sorbitol.
  Other Names: SPS
  Arms: Sodium Polystyrene Sulfonate
Drug: Silicified microcrystalline cellulose — Oral suspension in water of placebo administered three times (tid) daily for 48 hours.
  Other Names: Placebo
  Arms: Silicified microcrystalline cellulose

SUMMARY:
It is hypothesized that SPS is more effective than placebo control (alternative hypothesis) in lowering i-STAT potassium levels in subjects with i-STAT potassium levels between 5.0 - 6.5 mmol/l versus no difference between SPS and placebo control (null hypothesis).

DETAILED DESCRIPTION:
Subjects with mild to moderate hyperkalemia (i-STAT potassium levels between 5.0-6.5 mmol/l, inclusive) will be randomized 1:1 in a double-blind fashion to receive placebo or SPS (15g), administered tid with meals for 48 hours. Subjects will come back to the clinic on Study Day 9 for an End of Study (EOS) visit. Adverse experiences will be recorded.

Blood potassium levels will be evaluated by both i-STAT and the Local Laboratory prior to the first dose on Study Days 1 and 2, 1, 2, and 4 hours after the first dose on Study Day 1, 1 and 4 hours after the first dose on Study Day 2 and prior to breakfast on Study Day 3, after 48 hours of treatment.

Subjects who have i-STAT potassium levels > 6.5 mmol/l on Study Day 1 at the 4 hour post Dose 1 time point will be withdrawn from the study and will receive standard of care. If the i-STAT potassium value is between 6.1 and 6.5 mmol/l at the 4-hour post Dose 1 draw, subjects will be kept in the clinic for another 90 minutes post Dose 2 and another blood draw will be taken and an ECG will be performed. If the i-STAT potassium level is ≥ 6.2 mmol/l at this time point, the subject will be discontinued from the study and standard of care will be instituted. If the i-STAT potassium level is < 6.2 mmol/l, and the ECG does not show any of the ECG withdrawal criteria (see below), the subject will continue in the study.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent.
* Over 18 years of age.
* Mean i-STAT potassium values between 5.0 - 6.5 mmol/l inclusive, at screening (Study Day 0).
* Previous participation in Clinical ZS-002 or ZS-003 protocol(s). However, subjects cannot be enrolled in this study until at least 30 days have elapsed from their last dose in study ZS-003.
* Ability to have repeated blood draws or effective venous catheterization.
* Women of childbearing potential must be using two forms of medically acceptable contraception (at least one barrier method) and have a negative pregnancy test at screening.

Women who are surgically sterile or those who are post-menopausal for at least 2 years are not considered to be of child-bearing potential.

Exclusion Criteria:

* Pseudohyperkalemia signs and symptoms, such as excessive fist clenching hemolyzed blood specimen, severe leukocytosis or thrombocytosis.
* Subjects treated with lactulose, Xifaxan or other non-absorbed antibiotics for hyperammonemia within the last 7 days.
* Subjects treated with resins (such as Sevelamer acetate), calcium acetate, calcium carbonate, or lanthanum carbonate, within the last 7 days.
* Subjects treated with Sodium Polystyrene Sulfonate (SPS; e.g. Kayexalate®) or ZS (microporous, fractionated, protonated zirconium silicate) within the last 30 days.
* Subjects with a life expectancy of less than 3 months.
* Subjects who are HIV positive.
* Subjects who are severely physically or mentally incapacitated and who in the opinion of investigator are unable to perform the subjects' tasks associated with the protocol.
* Women who are pregnant, lactating, or planning to become pregnant.
* Subjects with diabetic ketoacidosis.
* Presence of any condition which, in the opinion of the investigator, places the subject at undue risk or potentially jeopardizes the quality of the data to be generated.
* Known hypersensitivity or previous anaphylaxis to ZS or to components thereof.
* Previous treatment with SPS.
* Treatment with a drug or device within the last 30 days that has not received regulatory approval at the time of study entry.
* Subjects with cardiac arrhythmias that require immediate treatment.
* Subjects on insulin where a stable dose has not yet been established.*
* Subjects on dialysis. * Subjects on stable insulin or insulin analogues can be enrolled. Subjects who have been on the same insulin dose and regimen for > 14 days are considered stable. Whenever possible, all blood draws collected prior to meals should be collected prior to insulin/insulin analogue treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Rasmussen, MD, Study Chair — ZS Pharma, Inc.
Locations (1):
- Riverside Clinical Research, Edgewater, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sodium Polystyrene Sulfonate: Oral suspension in water of 15g sodium polystyrene sulfonate administered three times (tid) daily for 48 hours without co-administration of Sorbitol.
  Enrollment: Assessed for eligibility (n= 36 )
  Excluded (n= 4)
  * Not meeting inclusion criteria (n= 4 )
  * Declined to participate (n= 0)
  * Other reasons (n= 0 )
  Randomized (n= 32 )
  Allocated to intervention (n= 15 ): ACTIVE
  * Received allocated intervention (n= 15)
  * Did not receive allocated intervention (give reasons) (n= 0 )
  Lost to follow-up (give reasons) (n= 0 )
  Discontinued intervention before study terminated (n= 1): non-serious adverse event
  Analyzed (n= 0)
  ◻ Excluded from analysis (give reasons) (n= 32 study terminated early due to safety reasons)
- Silicified Microcrystalline Cellulose: Oral suspension of placebo blended with pigment to have the same appearance, taste, odor and mode of administration as SPS.
  Enrollment: Assessed for eligibility (n= 36 )
  Excluded (n= 4)
  * Not meeting inclusion criteria (n= 4 )
  * Declined to participate (n= 0)
  * Other reasons (n= 0 )
  Randomized (n= 32 )
  Allocated to intervention (n= 17): PLACEBO
  * Received allocated intervention (n= 17 )
  * Did not receive allocated intervention (give reasons) (n= 0)
  Lost to follow-up (give reasons) (n= 0 )
  Analyzed (n= 0)
  ◻ Excluded from analysis (give reasons) (n= 32 study terminated early due to safety reasons)
Period: Overall Study
Arm/Group | Sodium Polystyrene Sulfonate | Silicified Microcrystalline Cellulose
Started | 15 | 17
Completed | 14 | 17
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Mean i-STAT serum potassium values between 5.0 - 6.5 mmol/l inclusive at screening (Study Day 0) plus meeting inclusion/exclusion eligibility criteria.
Groups:
- Sodium Polystyrene Sulfonate: Oral suspension in water of 15g sodium polystyrene sulfonate administered three times (tid) daily for 48 hours without co-administration of Sorbitol.
  Sodium polystyrene sulfonate (ACTIVE)
  Total Study Enrollment: Assessed for eligibility (n= 36 )
  Excluded (n= 4)
  * Not meeting inclusion criteria (n= 4 )
  * Declined to participate (n= 0)
  * Other reasons (n= 0 )
  Total Randomized (n= 32 )
  Allocated to intervention (n= 15 ): ACTIVE
  * Received allocated intervention (n= 15)
  * Did not receive allocated intervention (give reasons) (n= 0 )
  Lost to follow-up (give reasons) (n= 0 )
  Discontinued intervention before study terminated (n= 1): non-serious adverse event
  Analysed (n= 0)
  ◻ Excluded from analysis (give reasons) (n= 15): study terminated early due to safety reasons
- Silicified Microcrystalline Cellulose: Oral suspension of placebo blended with pigment to have the same appearance, taste, odor and mode of administration as SPS.
  Silicified microcrystalline cellulose (PLACEBO)
  Total Study Enrollment: Assessed for eligibility (n= 36 )
  Excluded (n= 4)
  * Not meeting inclusion criteria (n= 4 )
  * Declined to participate (n= 0)
  * Other reasons (n= 0 )
  Total Randomized (n= 32 )
  Allocated to intervention (n= 17): PLACEBO
  * Received allocated intervention (n= 17 )
  * Did not receive allocated intervention (give reasons) (n= 0)
  Lost to follow-up (give reasons) (n= 0 )
  Discontinued intervention (give reasons) (n= 0)
  Analysed (n= 0)
  ◻ Excluded from analysis (give reasons) (n= 17): study terminated early due to safety reasons
- Total: Total of all reporting groups
Arm/Group | Sodium Polystyrene Sulfonate | Silicified Microcrystalline Cellulose | Total
Number analyzed (Participants) | 15 | 17 | 32
Age, Continuous [Mean (Full Range); unit: years] | 71.1 [53 to 83] | 70.5 [50 to 88] | 70.8 [50 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Potassium Levels From Baseline After Administration of Sodium Polystyrene Sulfonate (SPS) Three Times a Day Without Co-administration of Sorbitol; Determine Incidence of Adverse Events.
Description: To perform a controlled evaluation of the safety and efficacy of 15g of SPS administered 3 times daily for 48 hours (6 doses) in patients with hyperkalemia (serum potassium levels between 5.0 - 6.5 mmol/l) at baseline.
Time Frame: First 48 hours
Population: Study prematurely terminated for safety reasons; no statistical analyses were conducted.
Groups:
- Sodium Polystyrene Sulfonate: Oral suspension in water of 15g sodium polystyrene sulfonate administered three times (tid) daily for 48 hours without co-administration of Sorbitol.
  Sodium polystyrene sulfonate
- Silicified Microcrystalline Cellulose: Oral suspension of placebo blended with pigment to have the same appearance, taste, odor and mode of administration as SPS.
  Silicified microcrystalline cellulose
Arm/Group | Sodium Polystyrene Sulfonate | Silicified Microcrystalline Cellulose
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Serum Sodium, Magnesium, Calcium Levels From Baseline After Administration of SPS.
Time Frame: First 48 hours
Population: Study was prematurely terminated for safety reasons; no statistical analyses were conducted.
Arm/Group | Sodium Polystyrene Sulfonate | Silicified Microcrystalline Cellulose
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Each study visit: Days 1, 2 and 9
Description: Participants were solicited for adverse events by systematic regular investigator assessment.
Groups:
- Sodium Polystyrene Sulfonate: Oral suspension in water of 15g sodium polystyrene sulfonate administered three times (tid) daily for 48 hours without co-administration of Sorbitol.
  Sodium polystyrene sulfonate (ACTIVE): Participants were solicited for adverse events at each study visit (i.e. Days 1, 2 and 9) by systematic regular investigator assessment.
- Silicified Microcrystalline Cellulose: Oral suspension of placebo blended with pigment to have the same appearance, taste, odor and mode of administration as SPS.
  Silicified microcrystalline cellulose (PLACEBO): Participants were solicited for adverse events at each study visit (i.e. Days 1, 2 and 9) by systematic regular investigator assessment.
Arm/Group | Sodium Polystyrene Sulfonate | Silicified Microcrystalline Cellulose
Serious Adverse Events (participants affected / at risk) | 2/15 | 0/17
Other Adverse Events (participants affected / at risk) | 7/15 | 3/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Polystyrene Sulfonate (N=15) | Silicified Microcrystalline Cellulose (N=17)
Prolonged QT Interval (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Polystyrene Sulfonate (N=15) | Silicified Microcrystalline Cellulose (N=17)
ST elevation (Cardiac disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (6) | 3 (3)
Flatulence (Gastrointestinal disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Stomach cramps (Gastrointestinal disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to the high frequency of adverse events in the SPS group, the independent Data Monitoring Committee (iDMC) recommended termination of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot publish any results related to the study without prior written approval of the Sponsor.